CLINICAL TRIAL: NCT02103985
Title: A Randomized, Open-Label, Two-Way Crossover Study to Determine the Effect of Food on the Pharmacokinetics of a Single JNJ-39823277 (TPI-1062) Dose in Healthy Male and Female Subjects
Brief Title: A Study of Effect of Food on the Pharmacokinetics of a Single JNJ-39823277 (TPI-1062) Dose in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR015718; TPI1062DEP1004 (Other: Johnson & Johnson Pharmaceutical Research and Development, L.L.C.)
Record Dates: First submitted 2014-04-01; First posted 2014-04-04 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
Keywords: Healthy; JNJ-39823277; JNJ-40917006; Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A (Experimental): Participants will receive 100 mg JNJ-39823277 under fed (after a high fat) condition.
  Interventions: Drug: JNJ-39823277
- Treatment B (Experimental): Participants will receive 100 mg JNJ-39823277 under fasted condition.
  Interventions: Drug: JNJ-39823277

INTERVENTIONS:
Drug: JNJ-39823277 — Participants will receive 100 mg of JNJ-39823277 tablet orally (by mouth) as a single dose.
  Other Names: TPI-1062

SUMMARY:
The purpose of this study is to evaluate the effect of food on the bioavailability of a single oral dose of JNJ-39823277 and its active metabolites.

DETAILED DESCRIPTION:
This is a randomized (the study medication is assigned by chance), open-label (all people know the identity of the intervention), single-center, 2 treatment-sequence, and crossover study (method used to switch participants from one treatment arm to another in a clinical study). The study consist of 3 phases: a screening phase (within 21 days before medication administration), a 2-period open-label treatment phase, during which each participant will receive 1 of 2 open-label treatment sequences, and the end-of-study or withdrawal assessments (within 7-11 days after the last dose of the study medication). Participants will be randomly assigned to 1 of 2 treatment-sequences: Treatment Sequence AB (dosing in fed [with high fat diet] condition followed by dosing in fasted [without food] condition) or Treatment Sequence BA (dosing in fasted condition followed by dosing in fed condition). Study medication administrations will be separated by a washout period (period when receiving no treatment) of 7 to 14 days. The study duration for each participant will be approximately 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be a healthy male or non-lactating healthy female
* Agrees to protocol-defined use of effective contraception
* If a woman, must have a negative serum ß-human chorionic gonadotropin (ß-hCG) pregnancy test at screening and on Day -1 of each treatment period
* Agree to abstain from all medication (except for allowed birth control), including prescription and non-prescription (including vitamins and natural or herbal remedies)

Exclusion Criteria:

* A history of clinically significant gastrointestinal, especially peptic ulcerations, gastrointestinal bleeding, ulcerative colitis, Crohn's disease or Irritable Bowel Syndrome, renal, hepatic, neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, psychiatric, especially those with a past history of depression, suicidal ideation or suicidal attempts, or cardiovascular disease
* Acute diarrhea or constipation in the 7 days before the predicted first study day. If screen occurs >7 days before first study day, this criterion will be determined on Day -1
* Participant has donated blood within 90 days or plasma within 30 days of study dosing
* Participant has used any over-the-counter or prescription medication, including vitamins, within 14 days prior to the study with the exception of acetaminophen
* Participant has consumed products containing grapefruit juice or grapefruit, Seville oranges (eg, orange marmalade), quinine (eg, tonic water), or xanthine (eg, chocolate, caffeine containing products) within 24 hours (72 hours in the case of grapefruit juice and Seville oranges) prior to start of study drug administration

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2009-05; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of JNJ-39823277 | Pre-dose; and 0.25, 0.50, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 30, 36 hours post-dose
  The Cmax is defined as maximum observed analyte concentration.
Time to Reach Maximum Observed Plasma Concentration (Tmax) of JNJ-39823277 | Pre-dose; and 0.25, 0.50, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 30, 36 hours post-dose
  The Tmax is defined as actual sampling time to reach maximum observed analyte concentration.
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of JNJ-39823277 | Pre-dose; and 0.25, 0.50, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 30, 36 hours post-dose
  The AUClast is area under the plasma concentration-time curve from time zero to the last quantifiable concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) of JNJ-39823277 | Pre-dose; and 0.25, 0.50, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 30, 36 hours post-dose
  The AUC(0-infinity) is area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of Area under Curve (AUC) last and C(last)/lambda(z), in which C(last) is the last observed quantifiable concentration.
Elimination Half-Life Period (T1/2) of JNJ-39823277 | Pre-dose; and 0.25, 0.50, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 30, 36 hours post-dose
  The T1/2 is the time measured for the plasma concentration to decrease by 1 half to its original concentration. It is associated with the terminal rate-constant (lambda[z]) of the semi logarithmic drug concentration-time curve, and is calculated as 0.693/lambda(z).
Maximum Observed Plasma Concentration (Cmax) of JNJ-40917006 (MC5 metabolite) | Pre-dose; and 0.25, 0.50, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 30, 36 hours post-dose
  The Cmax is defined as maximum observed analyte concentration.
Time to Reach Maximum Observed Plasma Concentration (Tmax) of JNJ-40917006 (MC5 metabolite) | Pre-dose; and 0.25, 0.50, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 30, 36 hours post-dose
  The Tmax is defined as actual sampling time to reach maximum observed analyte concentration.
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of JNJ-40917006 (MC5 metabolite) | Pre-dose; and 0.25, 0.50, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 30, 36 hours post-dose
  The AUClast is area under the plasma concentration-time curve from time zero to the last quantifiable concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) of JNJ-40917006 (MC5 metabolite) | Pre-dose; and 0.25, 0.50, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 30, 36 hours post-dose
  The AUC(0-infinity) is area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of Area under Curve (AUC) last and C(last)/lambda(z), in which C(last) is the last observed quantifiable concentration.
Elimination Half-Life Period (T1/2) of JNJ-40917006 (MC5 metabolite) | Pre-dose; and 0.25, 0.50, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 30, 36 hours post-dose
  The T1/2 is the time measured for the plasma concentration to decrease by 1 half to its original concentration. It is associated with the terminal rate-constant (lambda[z]) of the semi logarithmic drug concentration-time curve, and is calculated as 0.693/lambda(z).

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | Up to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research and Development, L.L C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (1):
- Lincoln, Nebraska, United States